CLINICAL TRIAL: NCT03368105
Title: Prevention of Clostridium Difficile Infections Using Lactobacillus Plantarum 299v Strain in Nephrology and Transplantation Department
Brief Title: Prevention of Clostridium Difficile Infections Using Lactobacillus Plantarum 299v Strain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SilesianMUKB-647/2017
Record Dates: First submitted 2017-12-04; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-09

CONDITIONS: Clostridium Difficile
Keywords: Clostridium difficile Infection; Lactobacillus plantarum 299v; organ transplantation; antibiotic-associated diarrhoea
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LP299v group (Experimental): Participants: one capsule of LP299v orally per a day during the entire period of antibiotic therapy.
  Interventions: Dietary Supplement: Prevention of C. difficile infections using LP299v strain
- Placebo group (Placebo Comparator): Participants: one capsule of placebo orally per a day during the entire period of antibiotic therapy.
  Interventions: Dietary Supplement: Prevention of C. difficile infections using LP299v strain

INTERVENTIONS:
Dietary Supplement: Prevention of C. difficile infections using LP299v strain — Patients treated with antibiotics and at high CDI risk (patients after organ transplantation or receiving immunosuppressive therapy for any other reason) will be enroll to study.
  We will divide participants into two group. Group 1 will receive one capsule of LP299v orally per a day during the entire period of antibiotic therapy. Group 2 will receive one capsule of placebo during the entire period of antibiotic therapy.

SUMMARY:
The aim of this study was to analyze whether the use of the LP299v strain reduces the risk of Clostridium difficile infection (CDI) among patients receiving antibiotics and hospitalized in the nephrology and transplantation ward.

Patients from risk group (receiving immunosuppressive drugs and treated with antibiotics) were enrolled into study.

Participants will be divided into two groups. First group will receive one capsule of Lactobacillus plantarum 299v (LP299v) orally per a day. Second group will receive placebo.

DETAILED DESCRIPTION:
Clostridium difficile is currently the most frequently identified pathogen causing antibiotic-associated diarrhoea and the main cause of nosocomial diarrhoea. In regard to observed worldwide increase rate of infection and mortality from CDI the prevention of Clostridium difficile infections seems to be crucial, especially in patients at CDI high risk. So far, it has not been unambiguously proven that probiotics are effective in the prevention of Clostridium difficile infection among patients undergoing antibiotic therapy.

The Lactobacillus plantarum 299v (LP299v) is a Gram-positive lactic acid bacteria that naturally occurs on the surface of human intestinal mucosa. Specific properties to the gut mucosa colonization are due to mannose-dependent adhesion of LP299v to the epithelium of human intestines.This ability of LP299v leads to reduction of bacterial translocation from the intestinal lumen into the blood vessels, can prevent adhesion of many pathogens to intestinal epithelium and modulate the inflammatory response of the epithelium. The strain 299v of Lactobacillus plantarum has been found to decrease the severity of gastrointestinal adverse effects during antibiotic therapy. Limited data are available regarding the efficacy of LP299v for preventing Clostridium difficile infections.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* organ transplantation or receiving immunosuppressive drugs for any other reasons
* antibiotics therapy

Exclusion Criteria:

* no consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Clostridium difficile infection | During hospitalization - average of 14 days

IPD SHARING:
Plan to Share IPD: Undecided